CLINICAL TRIAL: NCT03150797
Title: Melatonin for Adolescent Migraine Prevention Study (The MAP Study).
Brief Title: Melatonin for Adolescent Migraine Prevention Study
Acronym: MAP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Fund
Sponsor: Amy Gelfand (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Amy Gelfand, Director of Pediatric Headache UCSF Benioff Children's Hospital, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-19623
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Migraine
Keywords: UCSF; UCLA; melatonin; migraine; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Melatonin 3mg (Experimental): Melatonin 3mg
  Interventions: Drug: Melatonin
- Melatonin 6mg (Experimental): Melatonin 6mg
  Interventions: Drug: Melatonin
- Placebo oral capsule (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Melatonin — Melatonin
  Arms: Melatonin 3mg; Melatonin 6mg
Drug: Placebo oral capsule — Placebo
  Arms: Placebo oral capsule

SUMMARY:
This will be a randomized, multi-site double-blind placebo-controlled trial of melatonin (2 different dosing arms) vs. placebo for migraine prevention in adolescents. We intend to enroll approximately 210 participants over 15 months at two sites: UCLA and UCSF. The duration of participation for each participant will be 4 months.

DETAILED DESCRIPTION:
Participation includes 16 weeks of daily headache diary recording and taking the study pill every night, 1-2 hours before bed. Aside from the initial 1 hour enrollment visit, all remaining study procedures will be completed from home.

During the enrollment visit, history of migraine, questionnaires, a neurologic and physical exam (including weight, blood pressure, pulse, and respiratory rate) will be performed. Girls who have had their first period will undergo a urine pregnancy test and will be instructed to use birth control if they are sexually active.

For the first 8 week phase, participants will be instructed to take one study pill every night, 1-2 hours before bedtime and complete a daily headache diary from a smartphone. Phone call check-ins will occur at week 4 and week 8.

After the first 8 weeks of the study, participants who are eligible for the second phase of the study will be notified by study staff and will be sent the next set of study pills. Again, participants will be instructed to take the study pill every night, 1-2 hours before bedtime and complete a diary entry every evening.

Phone call check-ins will occur at week 12 and week 16. At the final 16 week phone call, additional questionnaires and study completion feedback will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-17-inclusive
2. Weight ≥40 kg, so as not to require mg/kg based dosing
3. Meets International Classification of Headache Disorders III beta1 criteria for migraine in children/adolescents (international standard diagnostic criteria for research)
4. Lives in the state of California- to allow shipping of study medication from our pharmacy
5. Has at least one parent who speaks English-in order to ensure good communication with study team by phone
6. Has daily access to a smartphone in order to provide daily headache diary data
7. A Parent/Guardian consents and the adolescent is cognitively capable of giving assent to participate
8. Either not on a migraine preventive medication, or if on one the dose has been stable for at least 4 weeks prior to enrollment, or are willing to wait to start the study until they have reached a stable dose for 4 weeks
9. Willing to not use OTC melatonin or change migraine preventives during the trial
10. Has ≥1 headache day per week, or 4-28 days of headache in a 28-day period Episodic headaches have been present for a minimum of 6 months-This lowers the likelihood of a secondary cause of headaches

Exclusion Criteria:

1. Continuous headache
2. History of seizures/epilepsy
3. Pregnant/lactating
4. Concomitant opioid or barbiturate overuse, wherein overuse is defined as ≥4 days per month of barbiturate containing compounds, ≥10 days per month of opioid containing compounds as these may impact sleepiness scales
5. If in the investigator's opinion there is a medical or psychiatric concern that makes them think the participant should not participate
6. Inability to swallow pills after teaching and practice History of nocturnal asthma, as evidenced by a having a diagnosis of asthma and symptoms that manifest as nighttime awakening due to cough, wheeze, and/or shortness of breath

Randomization Criteria:

1. Had 4-28 migraine/migrainous days in the 28-day period of weeks 5-8 of single-blind placebo treatment phase, but not continuous headache.
2. At least 80% compliance with headache diary (i.e. at least 23 headache diary days) during weeks 5-8 of single-blind placebo treatment phase.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Gelfand, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - UCLA Headache Research and Treatment Program, Los Angeles, California
  - University of California, San Francisco, (UCSF), San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Bigal ME, Lipton RB, Winner P, Reed ML, Diamond S, Stewart WF; AMPP advisory group. Migraine in adolescents: association with socioeconomic status and family history. Neurology. 2007 Jul 3;69(1):16-25. doi: 10.1212/01.wnl.0000265212.90735.64. PMID 17606878
- [Background] Arruda MA, Bigal ME. Migraine and migraine subtypes in preadolescent children: association with school performance. Neurology. 2012 Oct 30;79(18):1881-8. doi: 10.1212/WNL.0b013e318271f812. PMID 23109652
- [Background] Chang YS, Lin MH, Lee JH, Lee PL, Dai YS, Chu KH, Sun C, Lin YT, Wang LC, Yu HH, Yang YH, Chen CA, Wan KS, Chiang BL. Melatonin Supplementation for Children With Atopic Dermatitis and Sleep Disturbance: A Randomized Clinical Trial. JAMA Pediatr. 2016 Jan;170(1):35-42. doi: 10.1001/jamapediatrics.2015.3092. PMID 26569624
- [Background] Goncalves AL, Martini Ferreira A, Ribeiro RT, Zukerman E, Cipolla-Neto J, Peres MF. Randomised clinical trial comparing melatonin 3 mg, amitriptyline 25 mg and placebo for migraine prevention. J Neurol Neurosurg Psychiatry. 2016 Oct;87(10):1127-32. doi: 10.1136/jnnp-2016-313458. Epub 2016 May 10. PMID 27165014
- [Background] Masruha MR, de Souza Vieira DS, Minett TS, Cipolla-Neto J, Zukerman E, Vilanova LC, Peres MF. Low urinary 6-sulphatoxymelatonin concentrations in acute migraine. J Headache Pain. 2008 Aug;9(4):221-4. doi: 10.1007/s10194-008-0047-5. Epub 2008 Jul 2. PMID 18594760
- [Background] Masruha MR, Lin J, de Souza Vieira DS, Minett TS, Cipolla-Neto J, Zukerman E, Vilanova LC, Peres MF. Urinary 6-sulphatoxymelatonin levels are depressed in chronic migraine and several comorbidities. Headache. 2010 Mar;50(3):413-9. doi: 10.1111/j.1526-4610.2009.01547.x. Epub 2009 Oct 8. PMID 19817880
- [Background] Alstadhaug KB, Odeh F, Salvesen R, Bekkelund SI. Prophylaxis of migraine with melatonin: a randomized controlled trial. Neurology. 2010 Oct 26;75(17):1527-32. doi: 10.1212/WNL.0b013e3181f9618c. PMID 20975054
- [Background] Bougea A, Spantideas N, Lyras V, Avramidis T, Thomaidis T. Melatonin 4 mg as prophylactic therapy for primary headaches: a pilot study. Funct Neurol. 2016 Jan-Mar;31(1):33-7. doi: 10.11138/fneur/2016.31.1.033. PMID 27027892
- [Background] Fallah R, Shoroki FF, Ferdosian F. Safety and efficacy of melatonin in pediatric migraine prophylaxis. Curr Drug Saf. 2015;10(2):132-5. doi: 10.2174/1574886309666140605114614. PMID 24909684
- [Background] Miano S, Parisi P, Pelliccia A, Luchetti A, Paolino MC, Villa MP. Melatonin to prevent migraine or tension-type headache in children. Neurol Sci. 2008 Sep;29(4):285-7. doi: 10.1007/s10072-008-0983-5. Epub 2008 Sep 20. PMID 18810607
- [Background] Spilsbury JC, Drotar D, Rosen CL, Redline S. The Cleveland adolescent sleepiness questionnaire: a new measure to assess excessive daytime sleepiness in adolescents. J Clin Sleep Med. 2007 Oct 15;3(6):603-12. PMID 17993042

RESULTS

PARTICIPANT FLOW:
Period: Single-blind Placebo Run in Phase
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Started (In the single-blind phase, all participants started on placebo for 8 weeks. At the end of the 8 weeks, only those who had not dropped out and who met randomization criteria went on to the double-blind phase. Of the 59 who completed phase 1, only 44 met randomization criteria, of whom 42 were randomized (2 were not randomized due to error).) | 0 | 0 | 72
Completed | 0 | 0 | 59
Not Completed | 0 | 0 | 13
Period: Double Blind Phase
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Started (The reason this number does not match the number above is that in the single blind phase ALL participants received placebo.) | 14 | 14 | 14
Completed (i.e., provided at least 21/28 headache diary days during final four weeks of double-blind treatment (weeks 13-16 overall).) | 10 | 10 | 7
Not Completed | 4 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Enrolled in Single-blind Phase, But Did Not Randomize.: Placebo
  This group constitutes those who enrolled in the study and entered the single-blind phase, but did not go on to the double-blind randomized phase.
- Total: Total of all reporting groups
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule | Enrolled in Single-blind Phase, But Did Not Randomize. | Total
Number analyzed (Participants) | 14 | 14 | 14 | 30 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 14 | 14 | 30 | 72
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (2.1) | 14.3 (2.4) | 15.4 (1.5) | 14.4 (1.7) | 15.0 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 11 | 16 | 49
  Male | 4 | 2 | 3 | 14 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 1 | 0 | 0 | 1 | 2
  White | 9 | 10 | 9 | 20 | 48
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5 | 7 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 14 | 30 | 42

OUTCOME MEASURES:

1. Primary Outcome: Mean Migraine/Migrainous Days in Weeks 5-8 of Randomized Treatment Phase in Melatonin Treated Participants vs. Placebo.
Description: Mean migraine/migrainous days in weeks 5-8 of randomized treatment phase in melatonin treated participants vs. placebo. (Ultimately, as the data were not normally distributed, medians were more appropriate).
Time Frame: weeks 5-8 of randomized treatment phase
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 10 | 7
days | 2 [1 to 16] | 2 [0 to 6] | 2 [1 to 7]

2. Secondary Outcome: Mean Migraine/Migrainous Days in Weeks 5-8 of Randomized Treatment Phase in Melatonin 6 mg vs. Placebo.
Description: Mean migraine/migrainous days in weeks 5-8 of randomized treatment phase in melatonin 6 mg vs. placebo. (Medians reported when data were not normally distributed).
Time Frame: Weeks 5-8 of randomized treatment phase.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 10 | 7
days | 2 [1 to 16] | 2 [0 to 6] | 2 [1 to 7]

3. Secondary Outcome: Mean Migraine/Migrainous Days in Weeks 5-8 of Randomized Treatment Phase in Melatonin 3 mg vs. Placebo.
Description: Mean migraine/migrainous days in weeks 5-8 of randomized treatment phase in melatonin 3 mg vs. placebo.
Time Frame: Weeks 5-8 of randomized treatment phase.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 10 | 7
days | 2 [1 to 16] | 2 [0 to 6] | 2 [1 to 7]

4. Secondary Outcome: Mean Migraine/Migrainous Days in Weeks 5-8 of Randomized Treatment Phase in Melatonin 6 mg vs. Melatonin 3 mg.
Description: Mean migraine/migrainous days in weeks 5-8 of randomized treatment phase in melatonin 6 mg vs. melatonin 3 mg.
Time Frame: Weeks 5-8 of randomized treatment phase.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 10 | 7
days | 2 [1 to 16] | 2 [0 to 6] | 2 [1 to 7]

5. Secondary Outcome: Change in Mean Migraine/Migrainous Days From Weeks 5-8 of Single-blind Treatment Phase to Weeks 5-8 of Randomized Treatment Phase for Each Group.
Description: Change in mean migraine/migrainous days from weeks 5-8 of single-blind treatment phase to weeks 5-8 of randomized treatment phase for each group. (Medians reported when data were not normally distributed).
Time Frame: Weeks 5-8 of single-blind treatment phase to weeks 5-8 of randomized treatment phase.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 10 | 7
days | 2 [-1 to 7] | -1 [-3 to 0] | 0 [-5 to 3]

6. Secondary Outcome: Mean PedMIDAS (Pediatric Migraine Disability Assessment Score) in Weeks 5-8 of Randomized Treatment Phase in Each Melatonin Treated Group vs. Placebo, and in Each of the Three Pair-wise Group Comparisons.
Description: Mean PedMIDAS (headache related disability score) in weeks 5-8 of randomized treatment phase in each melatonin treated group vs. placebo, and in each of the three pair-wise group comparisons. PedMIDAS is a 6 question instrument for measuring headache related disability in children and adolescents.
Time Frame: Weeks 5-8 of randomized treatment phase.
Population: Data were not collected
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Mean CASQ (Cleveland Adolescent Sleepiness Questionnaire) Score in Weeks 5-8 of Randomized Treatment Phase in Melatonin Treated Group vs. Placebo, and in Each of the Three Pair-wise Group Comparisons.
Description: Mean CASQ score in weeks 5-8 of randomized treatment phase in melatonin treated group vs. placebo, and in each of the three pair-wise group comparisons. The CASQ is a 16-question instrument that uses Likert-like responses and has a score range from 16-80; higher scores indicate greater sleepiness
Time Frame: Weeks 5-8 of randomized treatment phase.
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 8 | 6
points | 33 (9) | 36 (6) | 28 (11)

8. Secondary Outcome: Number of Days Acute Medication is Used in Weeks 5-8 of Randomized Treatment Phase in Melatonin Treated Group vs. Placebo, and in Each of the Three Pair-wise Group Comparisons.
Description: Number of days acute medication is used in weeks 5-8 of randomized treatment phase in melatonin treated group vs. placebo, and in each of the three pair-wise group comparisons. This refers to the number of days that medication for the acute treatment of headache was used during the time frame.
Time Frame: Weeks 5-8 of randomized treatment phase.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 10 | 7
days | 5 [2 to 9] | 3 [0 to 5] | 3 [1 to 7]

9. Secondary Outcome: Number of Headache Days in Weeks 5-8 of Randomized Treatment Phase in Melatonin Treated Group vs. Placebo, and in Each of the Three Pair-wise Group Comparisons.
Description: Number of headache days in weeks 5-8 of randomized treatment phase in melatonin treated group vs. placebo, and in each of the three pair-wise group comparisons. This refers to number of headache days during the time period--regardless of whether they were migraine or not.
Time Frame: Weeks 5-8 of randomized treatment phase.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
Number analyzed (Participants) | 10 | 10 | 7
days | 8 [3 to 21] | 4 [1 to 11] | 5 [1 to 9]

ADVERSE EVENTS:
Time Frame: 8 week double-blind phase
Arm/Group | Melatonin 3mg | Melatonin 6mg | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/14 | 3/14 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin 3mg (N=14) | Melatonin 6mg (N=14) | Placebo Oral Capsule (N=14)
Headache worsening (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Headache worsening after head trauma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Worsened movement sensitivity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated heart rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Flu-like symptoms (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT03150797/Prot_SAP_000.pdf